CLINICAL TRIAL: NCT05795660
Title: The Effect of Platelet Rich Plasma for the Treatment of Osteochondral Lesions of the Talus: Randomized Controlled Trial
Brief Title: The Effect of Platelet Rich Plasma for the Treatment of Osteochondral Lesions of the Talus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Meshal Alhadhoud, Head of Orthopedic Surgery Department, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1736/2021
Record Dates: First submitted 2022-11-16; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Osteochondral Lesions of the Talus

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteochondral lesions of the talus group (Experimental): Patients will receive PRP injection.
  Interventions: Biological: platelet rich plasma
- Control group (Placebo Comparator): Patients will receive saline injection.
  Interventions: Biological: platelet rich plasma

INTERVENTIONS:
Biological: platelet rich plasma — platelet rich plasma injection
  Other Names: platelet rich plasma injection

SUMMARY:
Osteochondral lesion of the talus (OCL) results from the detachment of the talar cartilage which could also be associated with subchondral bone fragmentation due to trauma. OCL can be managed conservatively by immobilization and weight bearing restriction or surgically to stimulate the regeneration and the formation of fibrous cartilage including reparative or replacement approaches. OCL surgical intervention includes bone marrow stimulation or autologous osteochondral transplantation while the cartilage regeneration was found unsatisfactory with these interventions. However, introducing platelet rich plasma (PRP) as an adjacent intervention could enhance the cartilage regeneration in OCL due to the release of growth factors and bioactive components, which could in turn reduce the need for replacement interventions and improve the regeneration of the cartilage.

The literature was reviewed, and four randomized controlled trials have been found exploring the effect of PRP in OCL where both ankle function and pain were examined. The results of the previous studies have proved the effectiveness of PRP in managing OCL as an adjunct to microfracture surgery in improving ankle function and reducing pain which was superior to the surgical intervention alone and also superior to the injection of PRP alone. Despite the promising results, the previous studies were limited to several factors. There was a lack of blinding which could risk the results to expectation bias, and the follow up period was short in according to the MCMS, which is needed to monitor the long-term effect of the PRP and to document any potential adverse effects or relapse in the function. Additionally, all the previous studies performed blind injection. Additionally, the previous studies have not controlled the administration of analgesic which could risk the results of the pain effect.

The proposed study aims to examine the effect of PRP in the management of OCL using randomized double-blind control trial design to eliminate any expectation bias. Patients will be followed up for 12 months, and the PRP will be administered intra-operatively. Moreover, PRP concentration will be standardized. Analgesic will be controlled and documented as a confounded factor. Additionally, the quality of the repaired tissue and the regeneration of the hyaline cartilage will be examined using MRI at the end of the follow-up. Therefore, the study aims to examine the effectiveness of PRP in OCL using randomized controlled trial design.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of OCL, which will be confirmed with radiographs and magnetic resonance imaging.
* aged > or = 18 years < 60 year
* complain of ankle pain.

Exclusion Criteria:

* posterior OCL
* pregnancy
* ankle infection
* teroid injection within 6 months
* surgery of the involved joint with 6 months
* received glucosamine and/or chondroitin sulfate, or anticoagulant
* Systematic inflammatory condition
* substantial venous or lymphatic stasis in the legs
* Pathologies that my confound pain and functional assessment in the ankle (plantar fasciitis, Achilles tendonitis, sprains, and degenerative joint disease of the foot.
* Allergy to any of the component of the PRP injection, disabling degenerative joint disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle (AOFAS) score | 12 months

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request.